CLINICAL TRIAL: NCT03817840
Title: Novel Mediators of the Lipodystrophy and Metabolic Consequences of Cushing's Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: New York Obesity and Nutrition Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR7901
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cushing's Syndrome
Keywords: Glucocorticoids
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subjects will undergo 4mm punch biopsies of the SC, DC, and subcutaneous abdominal fat pads under local anesthesia (lidocaine). Biopsies will be performed by an interventional radiologist or surgeon. Specimens will be prepared for histologic analysis and for immunohistochemical analysis for brown and white adipose tissue markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment of Cushing's — Surgical resection of ACTH-secreting tumor to achieve cure of hypercortisolism
  Other Names: Medical treatment of hypercortisolism

SUMMARY:
This proposal will evaluate the glucocorticoid mediated changes in body fat distribution and metabolism that occur in patients with Cushing's disease. The objective is to identify the mechanisms that influence both the accumulation of lipodystrophic fat and also the changes in energy expenditure and metabolism that accompany them. The study is designed to determine if the high cortisol and AgRP levels in the blood of people living with Cushing's syndrome, either from taking steroid medications or from tumors, impact body fat and metabolism by turning off brown fat, which is a type of fat that increases one's metabolism.

DETAILED DESCRIPTION:
Cushing's disease (CD) is a disorder of chronic glucocorticoid (GC) excess that gives rise to a constellation of metabolic comorbidities and to a distinct lipodystrophic body habitus characterized by central adiposity, extremity wasting, and the accumulation of supraclavicular (SC) and dorsocervical (DC) fat in the region where human brown and beige adipose tissue is known to be concentrated. In spite of the recognized thermogenic capacity of select cervical adipocytes, the potential impact of lipomatous alterations in this depot on energy balance and metabolism in CD is unknown. To our knowledge, the "buffalo hump" and the supraclavicular fat pads - which are a sensitive physical finding for CD, have never been phenotypically characterized and the mechanisms underlying the GC mediated development of fat in these depots and the associated metabolic complications have not been explored in humans. The proposed research will advance our understanding of Cushing's lipodystrophy and its metabolic complications. Furthermore, it may lead to the identification of novel mediators and targetable pathways to attenuate the adverse effects of hypercortisolism on body composition and metabolism in CD, as well as in the significant population of patients treated with chronic GCs for an array of other clinical conditions. These findings may have important implications not only for those with Cushing's disease, but for the millions of Americans who are treated with chronic glucocorticoids for an array of clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 yrs
2. Body mass index (BMI) <35 kg/m2
3. Urine free cortisol (UFC) ≥150ug/d
4. Pituitary tumor >6mm on MRI or an inferior petrosal sinus sampling with central to peripheral plasma adrenocorticotropic hormone (ACTH) gradient
5. Normal renal and thyroid function
6. HbA1c ≤8.0.

Exclusion Criteria:

1. Smoking
2. Alcohol >2 drinks/day
3. Uncontrolled hypertension
4. HIV given potential for lipodystrophic confounding
5. Pregnancy and nursing
6. Use of beta-blockers, β-adrenergic or diabetes medications other than insulin
7. History of claustrophobia or difficulty lying flat
8. In-dwelling metal hardware.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACTH-dependent Cushing's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | Change from baseline REE at 3 months post-treatment
  Resting energy expenditure (REE) will be measured by whole room indirect calorimetry prior to and following cure of Cushing's Disease (CD).

SECONDARY OUTCOMES:
Total body adipose tissue volume | Change in total body adipose tissue volume from baseline at 3 months post-treatment
  Whole body MRI will be utilized to measure total body adipose tissue volume

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Page-Wilson, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Neuroendocrine Unit, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No